CLINICAL TRIAL: NCT02696876
Title: Safety and Efficacy of a Novel Synovium Brushing Method for Endogenous Mesenchymal Stem Cells Mobilisation During Knee Joint Microfracture for Cartilage Repair.
Brief Title: Synovium Brushing to Augmented Microfracture for Improved Cartilage Repair
Acronym: AURA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dennis McGonagle, Profession of Regenerative Medicine, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RR15/173
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Defect of Articular Cartilage; Cartilage Injury; Osteoarthritis, Knee
Keywords: Cartilage; Mesenchymal stromal cell; Microfracture; Knee; Defect; Injury; Stem cell; Autologous; Minimally manipulated
MeSH Terms: conditions — Osteoarthritis, Knee; Fractures, Stress; Wounds and Injuries | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Patients in this group will received conventional microfracture treatment as indicated for isolated cartilage defects and defined by the inclusion criteria.
  Interventions: Procedure: Microfracture
- Intervention group (Experimental): Patients in this group will also receive microfracture for the treatment of isolated cartilage defects in combination with arthroscopic synovial brushing to access and release synovial MSCs into the joint space.
  Interventions: Device: Arthroscopic synovial brushing

INTERVENTIONS:
Device: Arthroscopic synovial brushing — The specific and novel surgical procedure that will be carried out here is synovial membrane brushing using a novel device that has been shown to release MSCs from the synovium in vitro. This technique will be carried out in the setting of therapeutic microfracture for cartilage defects.
  Arms: Intervention group
Procedure: Microfracture — Microfracture or marrow-stimulation is a surgical procedure to repair small isolated cartilage defects by recruiting bone marrow mesenchymal stromal cells by creating small holes ('micro fractures') in the sub-chondral bone. These cells are entrapped in the ensuing blood clot and contribute to partial repair of the cartilage.
  Other Names: Marrow-stimulation
  Arms: Control group

SUMMARY:
This is a proof-of-concept study to determine the safety and efficacy of a novel device to increase the reparative capacity of the knee. The discovery of a resident population of mesenchymal stem cells (MSCs) within synovial fluid (SF) was the first description of this reparative cell population having direct access to superficial cartilage and joint structures. The ready access of SF MSC to cartilage and other joint tissues offers a novel strategy for joint repair. Current arthroscopic procedures result in the removal of all SF MSCs due to continuous irrigation throughout the procedure. The current study would benefit the patient by greatly increasing the reparative capacity of the joint by bolstering MSC numbers and retaining those MSCs within the joint after surgery. By accessing MSCs from the synovium it is anticipated that these cells would be entrapped/migrate into the marrow clot formed by microfracture of the sub-chondral bone. These MSCs would supplement those from the marrow and may result in faster, better quality repair.

DETAILED DESCRIPTION:
The synovium is a rich source of potent chondrogenic mesenchymal stromal cells (MSCs). Gaining access to this valuable source of regenerative cells could improve the outcome of joint restorative procedures. To avoid costly two-stage procedures and ex vivo manipulation, exploiting these autologous cells in a minimally invasive way with minimal manipulation could provide a novel cost-effective approach.

This study will evaluate the safety, feasibility and efficacy of a novel medical device (a synovial brush) and procedure (synovial brushing) to increase the number of autologous minimally manipulated MSCs in the knee. Twenty patients undergoing microfracture for isolated chondral defects will be randomly assigned to either a control group (microfracture only, 10 patients) or the intervention group (microfracture plus synovial brushing, 10 patients). The device is intended to increase the number of MSCs within the joint as a final stage during surgery, aiding repair by bolstering those MSCs recruited from the bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Isolated cartilage defects (<2cm2)
* Patients undergoing microfracture for repair of cartilage defects

Exclusion Criteria:

* Septic arthritis
* Infectious disease
* Revision joint surgery
* Meniscal damage requiring repair
* Ligament damage requiring repair
* Cartilage defect greater than 2cm2
* Contra-indications for MRI:

  * Pacemakers, Implantable Cardioverter defibrillators, implantable cardiac loop recorders
  * Surgical clips within the head
  * Certain inner ear implants
  * Neuro-electrical stimulators
  * Metal fragments within the eye or head

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01; Primary Completion 2023-01 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
The mean change in the number of MSCs present in the knee pre- and post- microfracture/microfracture plus arthroscopic synovial brushing. | 2 weeds

SECONDARY OUTCOMES:
Number of patients whose clinical effusion scores improve at 3, 6 and 12 months | 3, 6 and 12 months
Number of patients whose semi-quantitative MRI cartilage scores improve at 6 and 12 months | up to 12 months
Median KOOS scores at 3, 6 and 12 months (pain; other symptoms; function in daily living; function in sport; knee-related QoL; average score) | 3, 6 and 12 months
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 3, 6 and 12 months
  Median WOMAC scores at 3, 6 and 12 months (total; pain; stiffness; function)
Visual Analogue Scale (VAS) | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis G McGonagle, MB BcH BAO, Principal Investigator — University of Leeds
Locations (1):
- Chapel Allerton Orthopaedic Centre, Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No